CLINICAL TRIAL: NCT02046967
Title: Comparative Randomized Clinical Trial of Steam Ablation Versus Endovenous Laser Ablation for the Treatment of Great Saphenous Veins
Brief Title: Steam Ablation Versus Endovenous Laser Ablation for the Treatment of Great Saphenous Veins
Acronym: LAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, RR van den Bos, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ErasmusMC
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Varicose Veins; Varicose Veins of Leg With Long Saphenous Vein Distribution
Keywords: endovenous laser ablation; endovenous steam ablation; great saphenous veins; quality of life
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endovenous laser ablation (Active Comparator): Endovenous laser ablation with 940 nm bare fiber.
  Interventions: Procedure: Endovenous laser ablation with 940 nm bare fiber
- Endovenous steam ablation (Active Comparator): Endovenous steam ablation with steam vein sclerosis system.
  Interventions: Procedure: Endovenous steam ablation with steam vein sclerosis system.

INTERVENTIONS:
Procedure: Endovenous laser ablation with 940 nm bare fiber — Endovenous laser ablation with 940 nm Diode laser using a bare fiber for treating the Great Saphenous Vein.
  Other Names: EVLT; EVLA
  Arms: Endovenous laser ablation
Procedure: Endovenous steam ablation with steam vein sclerosis system. — Endovenous steam ablation with steam vein sclerosis.
  Other Names: SVS; EVSA
  Arms: Endovenous steam ablation

SUMMARY:
Endovenous laser ablation is a common therapy of great saphenous vein insufficiency with a very high success rate. It works by heating and thereby obliterating the vein. Steam ablation is a new therapy that also works by heating and thereby obliterating the vein. The hypothesis of this study is that steam ablation is as effective as laser ablation, but that it results in better secondary outcomes (e.g., lower pain scores).

DETAILED DESCRIPTION:
The study is a randomized clinical trial comparing two different therapies for endovenous ablation of great saphenous veins. The aim of the study is to test whether the anatomical success rate of Steam Ablation is not inferior to that of Endovenous laser ablation (EVLA) in treatment of great saphenous vein insufficiency and compare the treatment safety, patient reported outcomes and cost-effectiveness analyses between EVLA and Steam Ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Insufficiency of the GSV measured with ultrasound imaging, reflux > 0.5 s, and diameter of vein > 0.5 cm
* Symptoms of chronic venous insufficiency
* No prior treatment of the insufficient GSV
* Informed consent

Exclusion Criteria:

* Acute deep or superficial vein thrombosis
* Agenesis of deep vein system
* Vascular malformation or syndrome
* Post-thrombotic syndrome, occlusive type
* Pregnancy
* Immobility
* Allergy to lidocaine
* Arterial insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Obliteration of varicose vein and/ or absence of reflux (>0.5 sec. of retrograde flow over >10cm) along the treated segment of the great saphenous vein (GSV) at 12 and 52 weeks. | 52 weeks

SECONDARY OUTCOMES:
Major complications: deep and superficial venous thrombosis (embolic events), nerve injury, skin burns, and (sub)cutaneous infections. | 12 weeks
Minor complications: ecchymosis, pain and hyperpigmentation. | 12 weeks
Health related quality of life will be measured using the Dutch Translated Aberdeen Varicose Vein Questionnaire (AVVQ). | 12 weeks
Treatment satisfaction | 2 weeks
Pain score | 2 weeks
Venous Clinical Severity Score (VCSS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Renate R van den Bos, MD, PhD, Study Director — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Derived] van den Bos RR, Malskat WS, De Maeseneer MG, de Roos KP, Groeneweg DA, Kockaert MA, Neumann HA, Nijsten T. Randomized clinical trial of endovenous laser ablation versus steam ablation (LAST trial) for great saphenous varicose veins. Br J Surg. 2014 Aug;101(9):1077-83. doi: 10.1002/bjs.9580. Epub 2014 Jun 30. PMID 24981585